CLINICAL TRIAL: NCT00797433
Title: Outcomes of Mechanically Ventilated Patients With Low Serum Testosterone
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Khalid F. Almoosa, MD, University of Texas Health Science Center
Other Study IDs: GR-931
Record Dates: First submitted 2008-11-21; First posted 2008-11-25 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Acute Respiratory Failure
Keywords: testosterone; mechanical ventilation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mechanical ventilation: All male patients with acute respiratory failure requiring mechanical ventilation

SUMMARY:
This is a study to determine the testosterone serum levels in male patient with acute respiratory failure requiring mechanical ventilation. The objective is to determine if low levels exist in this population and if it correlates with length of mechanical ventilation.

Hypothesis: Serum testosterone levels in mechanically ventilated male patients are significantly decreased from normal levels and correlate with disease severity and outcomes.

DETAILED DESCRIPTION:
Study Objectives

1. To confirm and quantify the presence of hypotestosteronemia in critically ill male patients with acute respiratory failure requiring mechanical ventilation via endotracheal intubation.
2. To correlate serum testosterone levels with disease severity, short-term outcomes, and survival in mechanically ventilated male patients.
3. To determine if demographic patient characteristics, such as age, admitting diagnosis, or the presence of co-morbidities, affect serum testosterone levels during mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Age > 18
3. Admission diagnosis of acute respiratory failure requiring endotracheal intubation and mechanical ventilation for > 24 hours
4. APACHE II score > 15 (APACHE: Acute Physiology and Chronic Health Evaluation - general indicator of disease severity and outcomes predictor)

Exclusion Criteria:

1. Chronic mechanical ventilation (i.e. patients on mechanical ventilatory support for > 21 days for at least 6 hours per day)
2. Patients on mechanical ventilation for > 48 hours prior to MICU admission
3. Non-invasive mechanical ventilation
4. Patients intubated and mechanically ventilated for drug overdose and anticipated to be intubated for < 24 hours
5. Known diagnosis of hypogonadism (requiring testosterone hormonal supplementation) or currently receiving testosterone therapy or received testosterone therapy within 30 days of MICU admission
6. History of testicular, prostate or pituitary tumor
7. Chronic use of systemic steroids prior to admission
8. Terminally ill patients who are not expected to live longer that 3 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult male patients with acute respiratory failure on mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Serum testosterone level | Day 1, 3 and 7

SECONDARY OUTCOMES:
Length of mechanical ventilation | Days

CONTACTS AND LOCATIONS:
Overall Officials: Khalid F Almoosa, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States